CLINICAL TRIAL: NCT04185168
Title: Effects of Isoflavones on Hypertension, Serum Concentrations of Fructoseamine and Advanced Glycated End Products in Peritoneal Dialysis Patients
Brief Title: Isoflavones and Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, zahra yari, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Peritoneal Dialysis
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isoflavone (Active Comparator): 100 mg soy isoflavone (as 2 tablets)
  Interventions: Dietary Supplement: soy isoflavone
- control (Placebo Comparator): 2 tablets of placebo
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: soy isoflavone — 100 mg soy isoflavone (as 2 tablets)
  Arms: isoflavone
Other: control — 2 tablets of placebo
  Arms: control

SUMMARY:
The aim of this double-blind randomized clinical trial is to determine the effects of isoflavones on serum concentrations of fructoseamine and advanced glycated end products in peritoneal dialysis patients. Forty-four patients from shafa clinic will randomly assign to either isoflavone or placebo group. The patients in isoflavone group will receive 100 mg soy isoflavone (as 2 capsules) daily for 8 weeks, while the placebo group will receive identical placebo. At the baseline and the end of the study,7 ml blood will be collected from each patient after a 12-14-hours fasting and serum concentrations of fructoseamine, carboxymethyl lysine, pentosidine, glucose will be measured. Furthermore, blood pressure measurements will be performed twice with a ten-minute interval between testing

ELIGIBILITY:
Inclusion Criteria:

Continuous Ambulatory Peritoneal Dialysis for 6 months or more Body mass index below 35

Exclusion Criteria:

infections inflammatory diseases liver diseases Clinical diagnosis of cancer receiving glucocorticoid and anti-inflammatory drugs receiving isoflavone supplements Constant consumption of soy or foods containing soy in the diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-16 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
glucose | 8 weeks
  Serum concentrations of glucose
fructoseamine | 8 weeks
  Serum concentrations of fructoseamine
carboxymethyl lysine | 8 weeks
  Serum concentrations of carboxymethyl lysine
pentosidine | 8 weeks
  Serum concentrations of pentosidine
Systolic blood pressure | 8 weeks
  Systolic blood pressure
Diastolic blood pressure | 8 weeks
  Diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran (the Islamic Republic Of), Iran